CLINICAL TRIAL: NCT01405586
Title: Randomized Phase III Study of the Addition of Cisplatin in Combination With Gemcitabine as First-line Therapy for Elderly Patients With Advanced Non Small Cell Lung Cancer.
Brief Title: MILES-3: Cisplatin in Combination With Gemcitabine for Elderly Patients With Lung Cancer
Acronym: MILES-3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MILES-3; 2009-013540-36 (EudraCT Number)
Record Dates: First submitted 2010-02-26; First posted 2011-07-29 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Stage IIIB
Keywords: elderly; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gemcitabine (Active Comparator)
  Interventions: Drug: Gemcitabine
- gemcitabine + cisplatin (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 days 1 and 8 every 3 weeks for 6 cycles
  Arms: gemcitabine + cisplatin
Drug: Gemcitabine — 1200 mg/m2 days 1 and 8 every 3 weeks for 6 cycles
  Arms: gemcitabine
Drug: Cisplatin — 60 mg/m2 day 1 every 3 weeks for 6 cycles
  Arms: gemcitabine + cisplatin

SUMMARY:
The purpose of this study is to evaluate the addition of cisplatin to first-line chemotherapy with gemcitabine in elderly patients with non small cell lung cancer in terms of overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological diagnosis of non small-cell lung cancer (NSCLC)
* Stage III B or Stage IV disease
* Age > or = 70 years
* ECOG Performance status 0 or 1
* Patient at first diagnosis or with recurrence after primary surgery
* At least one target or non-target lesion according to RECIST criteria
* Life expectancy of at least 3 months
* Neutrophils > 1500/mm3, platelets > 100,000/mm3, hemoglobin > 10g/dl
* Creatinine < 1.5 x the upper normal limit
* AST and ALT < 2.5 x the upper normal limits (< 5 x the upper normal limit in the presence of hepatic metastasis)
* Bilirubin < 1.5 x the upper normal limit
* Signed informed consent

Exclusion Criteria:

* Previous chemotherapy for advanced disease
* History of malignant neoplasm within the previous 5 years (not including non-melanoma skin carcinoma and in-situ carcinoma of the uterine cervix, provided they are being adequately treated)
* Symptomatic cerebral or spinal cord metastasis
* Myocardial infarct within the last 12 months
* Systemic disease not controlled with treatment (active infection, cardiovascular, hepatic, renal or metabolic) that would not, in the opinion of the investigator, permit the patient to undergo chemotherapy.
* Known or suspected hypersensitivity to any of the drugs used in the study
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or give informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 299 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
overall survival | one year

SECONDARY OUTCOMES:
worst grade toxicity per patient | at end of each 3 week cycle of chemotherapy
  worst toxicity per patient according to Common Toxicitity Criteria for Adverse Events v. 4.03
progression free survival | every 9 weeks
quality of life | baseline and 8, 21, 29, and 42 days after therapy initiated
objective response | after 9 and 18 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hopital, Avellino, Italy, Division of Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics
Locations (49):
- Italy (49):
  - Ospedale Villa Scassi, Genova, GE
  - Policlinico Giaccone, Palermo, PA
  - Azienda Ospedaliera Universitaria Senese, Siena, SI
  - Ospedale San Lazzaro, Alba
  - Ospedale Regina Apostolorum, Albano Laziale
  - AOU Ospedale Riuniti Umberto I, Ancona
  - ASL Latina Distretto 1 Aprilia Univ.degli Studi di Roma, Aprilia
  - Ospedale Cardinale Massaia, Asti
  - S. Giuseppe Moscati, Avellino
  - Centro Riferimento Oncologico, Aviano
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Ospedale A. Cardarelli, Campobasso
  - Ospedale Ramazzini di Carpi, Carpi
  - Ospedale S. Spirito, Casale Monferrato
  - A.O. Garibaldi Nesima, Catania
  - Ospedale Mater Domini, Catanzaro
  - Ospedale della Madonna della Navicella, Chioggia
  - Ospedale Civile di Faenza, Faenza
  - A.O.U. Arcispedale Sant'Anna di Ferrara, Ferrara
  - Ospedale Don Luigi Di Liegro, Gaeta
  - IRCCS San Martino -IST Genova, Genova
  - Ospedale F. Veneziale, Isernia
  - A.O. Vito Fazzi-Lorusso, Lecce
  - Ospedale Civile di Legnano, Legnano
  - Istituto Sceintifico Romagnolo, Meldola
  - Ospedale L. Sacco Polo Universitario, Milan
  - Ospedale San Paolo, Milan
  - U.L.S.S. 13, Mirano
  - Ospedale San Gerardo, Monza
  - Azienda Ospedaliera Cardarelli, Napoli
  - Second University of Naples, Napoli
  - A.O. Università Federico II, Napoli
  - AORN Ospedale dei Colli - Osp Monaldi, Napoli
  - Istituto Nazionale dei Tumori, Napoli
  - Istituto Oncologico Veneto, Padua
  - Ospedale Andrea Tortora Pagani - Ospedale Civile Umbero I, Pagani
  - Casa di Cura La Maddalena, Palermo
  - Ospedale Buccheri La Ferla - Fatebenefratelli, Palermo
  - Fondazione Salvatore Maugeri, Pavia
  - Ospedale Guglielmo d Saliceto-Piacenza, Piacenza
  - Azienda Ospedaliera S. Carlo, Potenza
  - Ospedale S. Maria delle Croci, Ravenna
  - Ospedale Umberto I, Ravenna
  - A.O. S. Camillo Forlanini, Roma
  - Campus Biomedico Policlinio Universitario, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma
  - Ospedale S. Andrea, Vercelli
  - Ospedale S. Bortolo ULSS 6, Vicenza
  - ASL Viterbo - Ospedale Belcolle, Viterbo